CLINICAL TRIAL: NCT05553314
Title: Slow-release CArvedilol in Patients With REduced Strain and Preserved Ejection Fraction Heart Failure (CARE-preserved HF): A Prospective Randomized, Double-Blinded, Multicenter Study
Brief Title: Carvedilol in HF With Preserved EF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Samsung Medical Center (Other); Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARE-preserved HF
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Beta Blocker; Myocardial Strain
Keywords: HFPEF; beta-blocker; reduced strain; BNP
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double-blinded, placebo-controlled study
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol-group (Experimental): Patients receiving carvedilol
  Interventions: Drug: Carvedilol
- Placebo-group (Placebo Comparator): Patients receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — patients randomized to carvedilol group will receive carvedilol-SR.
  Other Names: carvedilol slow-release (SR)
  Arms: Carvedilol-group
Drug: Placebo — patients randomized to placebo group will receive placebo.
  Arms: Placebo-group

SUMMARY:
Beta-blockers improve clinical outcomes in heart failure and reduced ejection fraction (HFrEF); but not in those with preserved EF. Global longitudinal strain (GLS) is a prognostic factor independent of left ventricular ejection fraction (LVEF). In a retrospective with 1969 patients with HF and LVEF of ≥40%, beta-blocker was associated with improved survival in those with low GLS (GLS <14%), but not in those with GLS ≥14%. In this prospective, randomized clinical study, the investigators will assess the effect of slow-release carvedilol in patients with HFpEF and hypertension. The primary endpoint is the time-averaged proportional changes in NT-proBNP level and GLS change from baseline to month 6.

ELIGIBILITY:
Inclusion Criteria:

* age ≥20 yrs
* symptomatic HFpEF with LVEF≥50%
* NT-proBNP ≥220 pg/ml (sinus rhythm) or ≥660 pg/ml(AF) (BNP ≥80 pg/ml (sinus rhythm) or ≥240 pg/ml(AF) )
* SBP≥140mmHg and/or DBP ≥90mmHg, or if taking anti-hypertensive medication, SBP ≥110mmHg.
* LAVI≥29(sinus rhythm)/34ml/m2 (AF) or LVMI≥115(male)/95(female) g/m2
* meet one the following

  1. Average E/e'≥ 9
  2. Septal e' < 7 cm/s
  3. Lateral e' <10 cm/s
  4. TR velocity > 2.8 m/s
  5. PASP > 35 mmHg
  6. GLS < 16%

Exclusion Criteria:

* systolic blood pressure < 110 mmHg, or heart rate < 60 beats/min
* contra-indication to beta-blockers
* creatinine> 2.4mg/dL
* amyloidosis, hypertrophic cardiomyopathy with obstruction, severe aortic or mitral valve disease, acute coronary syndrome, Cerebrovascular event within 6 months, PCI within 3 months before
* AST/ALT >3 x normal upper range

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP change | 6 months
  Time averaged NT-proBNP change from baseline to 6 months
GLS change | 6 months
  Change of GLS from baselin to 6 months

SECONDARY OUTCOMES:
off-level NT-proBNP | 6 months
  Decrease in NT-proBNP > 10% from baseline to 6 months
Mortality | 6 months
  All-cause mortality from baseline to 6 months
rehospitalization | 6 months
  rehospitalization from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, MD, PhD, Principal Investigator — Seoul National Univeristy Bundang Hospital
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Il-won
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park JJ, Park JB, Park JH, Cho GY. Global Longitudinal Strain to Predict Mortality in Patients With Acute Heart Failure. J Am Coll Cardiol. 2018 May 8;71(18):1947-1957. doi: 10.1016/j.jacc.2018.02.064. PMID 29724346
- [Result] Yamamoto K, Origasa H, Hori M; J-DHF Investigators. Effects of carvedilol on heart failure with preserved ejection fraction: the Japanese Diastolic Heart Failure Study (J-DHF). Eur J Heart Fail. 2013 Jan;15(1):110-8. doi: 10.1093/eurjhf/hfs141. Epub 2012 Sep 14. PMID 22983988
- [Result] Park JJ, Choi HM, Hwang IC, Park JB, Park JH, Cho GY. Myocardial Strain for Identification of beta-Blocker Responders in Heart Failure with Preserved Ejection Fraction. J Am Soc Echocardiogr. 2019 Nov;32(11):1462-1469.e8. doi: 10.1016/j.echo.2019.06.017. Epub 2019 Sep 17. PMID 31540679
- [Derived] Yoon M, Park SJ, Yoo BS, Choi DJ. The effect of sustained-release CARvedilol in patients with hypErtension and heart failure with preserved ejection fraction: a study protocol for a pilot randomized controlled trial (CARE-preserved HF). Front Cardiovasc Med. 2024 Apr 26;11:1375003. doi: 10.3389/fcvm.2024.1375003. eCollection 2024. PMID 38737708